CLINICAL TRIAL: NCT06572176
Title: Investigation of Fluorescent Concretization Intervention on Intensive Care Nurses' Hand Hygiene Training According to the Kirkpatrick Model: A Randomised Controlled Study
Brief Title: Investigation of Fluorescent Concretization Intervention on Intensive Care Nurses' Hand Hygiene Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hulya Yilmaz, Assistant Professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-7/18
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Hand; Health Care Associated Infection; Training Group, Sensitivity
Keywords: health care associated infections; fluorescent; hygiene; intensive care units
MeSH Terms: conditions — Cross Infection; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: A cluster-randomized controlled pretest-posttest and follow-up research design were used.
Masking Description: Because of the nature of the device and the procedure of fluorescent, blinding couldn't be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: With fluorescent concretization group (Experimental): Nurses were given the fluorescent lotion and asked to apply it all over their hands. The CE-certified test lotion is in gel form and is safety-approved. The lotion disperses particles the same size as bacteria on the skin. These particles settle on the skin, similar to the behavior of microorganisms, but disappear with hand washing under the influence of fluorescent light. They were then asked to wash their hands with 4 ml of soap. Two researchers marked the hand washing steps independently using the "Hand Washing Skill Checklist." The duration of hand washing was recorded with a mobile stopwatch for each participant. Hand washing efficiency was evaluated using the "Derma Litecheck" device. UV rays were used after using the test lotion and drying the hands. Since any fluorescent material left on the hands would shine under UV light, it was possible to judge how well the hands were cleansed. The dirty spots were shown to the participants, and the reason for this was discussed.
  Interventions: Behavioral: With fluorescent concretization group
- Control: Without fluorescent concretization group (No Intervention): The same interventions were repeated without fluorescent concretization and UV-A light intervention.

INTERVENTIONS:
Behavioral: With fluorescent concretization group — Nurses were given the fluorescent lotion and asked to apply it all over their hands. The CE-certified test lotion is in gel form and is safety-approved. The lotion disperses particles the same size as bacteria on the skin. These particles settle on the skin, similar to the behavior of microorganisms, but disappear with hand washing under the influence of fluorescent light. They were then asked to wash their hands with 4 ml of soap. Two researchers marked the hand washing steps independently using the "Hand Washing Skill Checklist." The duration of hand washing was recorded with a mobile stopwatch for each participant. Hand washing efficiency was evaluated using the "Derma Litecheck" device. UV rays were used after using the test lotion and drying the hands. Since any fluorescent material left on the hands would shine under UV light, it was possible to judge how well the hands were cleansed. The dirty spots were shown to the participants, and the reason for this was discussed.
  Other Names: fluorescent concretization group
  Arms: Experimental: With fluorescent concretization group

SUMMARY:
Aim: The primary objective was to assess the effect of fluorescent concretization intervention on intensive care nurses' hand-washing efficiency, skill performance, and duration scores during the training process. A secondary objective was to investigate the intensive care nurses to determine their level of hand hygiene knowledge before and after the training.

Design: Cluster-randomised controlled pretest-posttest and follow-up research design was used.

Methods: This study was conducted at a tertiary hospital in XX province, Türkiye. Seventy-six nurses from intensive care units participated in hand hygiene training. In addition to routine hand hygiene training, the participants in the intervention group (n=39) had their hand washing efficiency evaluated using ultraviolet A light. The dirty spots were shown to the participants, and the reasons were discussed. The participants in the control group (n=37) received hand washing training without fluorescent concretization and ultraviolet light intervention. The Hand Hygiene theoretical information is an evidence-based workplace intervention delivered by trained facilitators across two training. Hand Hygiene Information Forms were administered upon registration and before randomisation of all participants immediately after the final training. Two independent researchers observed Hand Washing Skill Checklist and Efficacy forms in three follow-ups (before training, 15 days after training, and four months after training).

DETAILED DESCRIPTION:
Aim: Nurses have a pivotal role in preventing and managing healthcare-acquired/associated infections by effective hand washing. The primary objective was to assess the effect of fluorescent concretization intervention on intensive care nurses' hand-washing efficiency, skill performance, and duration scores during the training process. A secondary objective was to investigate the intensive care nurses to determine their level of hand hygiene knowledge before and after the training.

Design: Cluster-randomised controlled pretest-posttest and follow-up research design was used.

Methods: This study was conducted at a tertiary hospital in XX province, Türkiye. Seventy-six nurses from intensive care units participated in hand hygiene training. In addition to routine hand hygiene training, the participants in the intervention group (n=39) had their hand washing efficiency evaluated using ultraviolet A light. The dirty spots were shown to the participants, and the reasons were discussed. The participants in the control group (n=37) received hand washing training without fluorescent concretization and ultraviolet light intervention. The Hand Hygiene theoretical information is an evidence-based workplace intervention delivered by trained facilitators across two training. Hand Hygiene Information Forms were administered upon registration and before randomisation of all participants immediately after the final training. Two independent researchers observed Hand Washing Skill Checklist and Efficacy forms in three follow-ups (before training, 15 days after training, and four months after training).

ELIGIBILITY:
Inclusion Criteria:

* nurses who have not received previous training on UVA-supported hand hygiene devices
* nurses who have not visibly damaged skin integrity on the hands
* Nurses are willing to participate in the study and take primary responsibility for patient care.
* nurses who have six months or more of intensive care experience

Exclusion Criteria:

* nurses who have received previous training on UVA-supported hand hygiene devices.
* nurses who do not have visibly damaged skin integrity on the hands.
* Nurses are willing to participate in the study and take primary responsibility for patient care.
* nurses who have six months or less of intensive care experience

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Hand Washing Skill Efficacy (HWSE) | through study completion, an average 1 year
  The hands were examined in seven areas: the palm, the back of the hand, and between the fingers, specifically the thumb, fingertips, nails, the anterior side of the wrist, and the posterior side. Under the UV light, dirty spots were marked separately for the right and left hands. The dirty spot was calculated as 1 point, and the clean spot was calculated as 0 points. 0-3-point range was considered clean; 4-7 point range was considered dirty (Škodová et al., 2015). ICC coefficient was 0.98 for the right HWSE before training, 1.0 after 15 days, and 1.0 at four months after training. The ICC coefficient was 0.96 for the left HWSE before training, 1.0 at 15 days after training, and 1.0 at four months after training. Two independent researchers completed this form in three repeated follow-ups.

SECONDARY OUTCOMES:
Hand Hygiene Information Form (HHIF) | through study completion, an average 1 year
  The form was prepared in line with the literature to determine participants' socio-demographic characteristics and knowledge of hand hygiene. In line with the training content, the items in the information form consisted of the history of hand hygiene, transmission of microorganisms, bacterial flora, glove use, surgical hand washing and scrubbing, hand hygiene products, hand hygiene compliance, and HAIs. The HHIF items created by the research team were presented to experts (n=10), including an assessment and measurement expert. As a result of expert evaluations, the Content Validity Index (CVI) was calculated as 1.0. Items with low CVI were excluded. Then, "HHIF" and "Hand Hygiene Training Guide for Intensive Care Nurses" were finalized after the pilot application with five intensive care nurses outside the study group. The form consisted of 19 items on HH topics. The lowest and highest scores that can be obtained from the form were 0 and 100, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya YILMAZ, Phd, Msc, Principal Investigator — Bursa Uludag University, Faculty of Health Sciences; Dilan Ayhan, Msc, Study Chair — Health Research and Application Center, Faculty of Medicine, Bursa Uludag University; Dilek YILMAZ, Phd, Msc, Study Chair — Bursa Uludag University, Faculty of Health Sciences; Yılmaz Özen, Professor, Study Chair — Health Research and Application Center, Faculty of Medicine, Bursa Uludag University
Locations (1):
- Bursa Uludag University Health Sciences Faculty of the Nursing Department, Nilufer, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Concept: H.Y., D.A., D.Y., Y.Ö. Design: H.Y., D.A., D.Y., Y.Ö. Supervision: H.Y., D.A., D.Y., Y.Ö. Materials: H.Y., D.A., D.Y., Y.Ö. Data Collection and/or Processing: H.Y., D.A. Analysis and/or Interpretation: Statistician. Literature Search: H.Y., D.A., D.Y., Y.Ö. Writing: H.Y. Critical Reviews: D.A., D.Y.

REFERENCES:
- [Background] Bounou L, Katelani S, Panagiotopoulou KI, Skouloudaki AI, Spyrou V, Orfanos P, Lagiou P. Hand hygiene education of Greek medical and nursing students: A cross-sectional study. Nurse Educ Pract. 2021 Jul;54:103130. doi: 10.1016/j.nepr.2021.103130. Epub 2021 Jun 28. PMID 34246184
- [Background] Cambil-Martin J, Fernandez-Prada M, Gonzalez-Cabrera J, Rodriguez-Lopez C, Almaraz-Gomez A, Lana-Perez A, Bueno-Cavanillas A. Comparison of knowledge, attitudes and hand hygiene behavioral intention in medical and nursing students. J Prev Med Hyg. 2020 Apr 2;61(1):E9-E14. doi: 10.15167/2421-4248/jpmh2020.61.1.741. eCollection 2020 Mar. PMID 32490263
- [Background] Diefenbacher S, Fliss PM, Tatzel J, Wenk J, Keller J. A quasi-randomized controlled before-after study using performance feedback and goal setting as elements of hand hygiene promotion. J Hosp Infect. 2019 Apr;101(4):399-407. doi: 10.1016/j.jhin.2019.02.001. Epub 2019 Feb 8. PMID 30738912
- [Background] Du Q, Zhang D, Hu W, Li X, Xia Q, Wen T, Jia H. Nosocomial infection of COVID-19: A new challenge for healthcare professionals (Review). Int J Mol Med. 2021 Apr;47(4):31. doi: 10.3892/ijmm.2021.4864. Epub 2021 Feb 4. PMID 33537803
- [Derived] Yilmaz H, Ayhan D, Yilmaz D, Ozen Y. Investigation of Fluorescent Concretisation Intervention on Intensive Care Nurses' Hand Hygiene Training According to the Kirkpatrick Model: A Cluster Randomised Controlled Study. Nurs Crit Care. 2025 Sep;30(5):e70141. doi: 10.1111/nicc.70141. PMID 40814898